CLINICAL TRIAL: NCT06192433
Title: Repeated Transcranial Magnetic Stimulation in the Elderly With Cognitive
Brief Title: Repeated Transcranial Magnetic Stimulation in the Elderly With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202314
Record Dates: First submitted 2023-10-13; First posted 2024-01-05 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Dementia; Cognitive Impairment, Mild
Keywords: high-frequency transcranial magnetic stimulation; cognitive impairment; Dementia
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This study is a Randomized Controlled Trial designed to investigate the effects of different frequencies of transcranial magnetic stimulation (TMS) as non-pharmacological treatment for patients with mild cognitive impairment or dementia. The trial employs a Parallel Study Design, where two groups of participants are treated concurrently with either high-frequency transcranial magnetic stimulation (40 Hz rTMS) or moderately high-frequency transcranial magnetic stimulation (10 Hz rTMS).
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants: Participants are masked or blinded to their group assignment. This blinding is implemented to reduce potential bias in the study, as participants are unaware of the treatment they receive.
  Assessors: The individuals who perform the cognitive function assessments are also blinded to the group assignment of the participants. They do not know whether a participant belongs to the high-frequency group (40Hz) or the moderately high-frequency group (10Hz). This dual blinding, of both participants and assessors, is important to ensure the integrity and validity of the study's results."
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-frequency repetitive transcranial magnetic stimulation group (40Hz) (Experimental): High-Frequency Group (40Hz): Participants in this arm receive high-frequency transcranial magnetic stimulation (rTMS) at 40Hz for a specified duration and intensity on the bilateral dorsolateral prefrontal cortex (DLPFC). The stimulation parameters and rest periods are outlined in the study description.
  Interventions: Device: High-frequency repetitive transcranial magnetic stimulation (40Hz)
- Moderately high-frequency repetitive transcranial magnetic stimulation group (10Hz) (Active Comparator): Moderately High-Frequency Group (10Hz): Participants in this arm receive moderately high-frequency transcranial magnetic stimulation (TMS) at 10Hz for a specified duration and intensity on the bilateral dorsolateral prefrontal cortex (DLPFC). The stimulation parameters and rest periods are outlined in the study description.
  Interventions: Device: Moderately high-frequency repetitive transcranial magnetic stimulation (10Hz)

INTERVENTIONS:
Device: High-frequency repetitive transcranial magnetic stimulation (40Hz) — Participants in this group receive high-frequency TMS at 40 Hz. The TMS intervention is applied to the bilateral dorsolateral prefrontal cortex (DLPFC). Each patient undergoes this TMS treatment for a course of 10 consecutive working days. The specific parameters for TMS include pulses at 40 Hz with an intensity set at 40% of the maximum intensity. Each pulse lasts for 2 seconds, followed by a 58-second rest period. On each treatment day, patients receive 30 sets of stimulation, with 15 stimulations applied to the left side and 15 to the right side, totaling 2400 pulses.
  Arms: High-frequency repetitive transcranial magnetic stimulation group (40Hz)
Device: Moderately high-frequency repetitive transcranial magnetic stimulation (10Hz) — Participants in this group receive moderately high-frequency TMS at 10 Hz. Similar to the high-frequency group, the TMS intervention targets the bilateral dorsolateral prefrontal cortex (DLPFC) and is administered for a course of 10 consecutive working days. The TMS parameters for this group involve pulses at 10 Hz with an intensity set at 90% of the maximum intensity. Each pulse lasts for 4 seconds, followed by a 56-second rest period. As in the high-frequency group, patients in this group also receive 30 sets of stimulation per treatment day, with 15 stimulations applied to the left side and 15 to the right side, totaling 2400 pulses.
  Arms: Moderately high-frequency repetitive transcranial magnetic stimulation group (10Hz)

SUMMARY:
Introduction and Purpose:

In recent years, non-pharmacological treatment methods for dementia patients have been gradually explored. Among these, Transcranial Magnetic Stimulation (TMS) has been proposed as a non-invasive treatment option. However, the optimal frequency and stimulation site for repetitive transcranial magnetic stimulation have not been definitively determined.

Methods:

This study is a randomized controlled trial. We randomly assigned 30 patients with mild cognitive impairment or dementia to the high-frequency transcranial magnetic stimulation group (40 Hz rTMS) or the moderately high-frequency transcranial magnetic stimulation group (10 Hz rTMS). Stimulation was applied to the bilateral dorsolateral prefrontal cortex (DLPFC). Each patient received a course of treatment for 10 consecutive working days. The high-frequency group received pulses at 40 Hz with an intensity of 40% of the maximum intensity for 2 seconds followed by a 58-second rest period, per set. The moderately high-frequency group received pulses at 10 Hz with an intensity of 90% of the maximum intensity for 4 seconds followed by a 56-second rest period, per set. Each day, patients received 30 sets of stimulation (15 times on the left side and 15 times on the right side), totaling 2400 pulses. Cognitive assessments were conducted on patients before and after the treatment course. Quantitative analysis will be performed using the Statistical Package for the Social Sciences statistical software. The Kolmogorov-Smirnov test will be used to check if the data follows a normal distribution. The chi-squared test will compare differences in baseline categorical variables between the groups, while independent t-tests or the Mann-Whitney U Test will compare baseline differences in continuous variables to assess the effectiveness of random assignment. Analysis of variance (ANOVA) and post-hoc comparisons will be used to compare intergroup and intragroup differences. The significance level is set at α = 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 and above.
2. Have received at least 2 years of education.
3. Diagnosed with dementia or Mild Cognitive Impairment (MCI).
4. Clinical Dementia Rating (CDR) score of ≥0.5.

Exclusion Criteria:

1. Mental illness.
2. Alcohol or substance addiction.
3. History of heart rhythm disorders.
4. History of epilepsy.
5. History of brain injury.
6. Underwent neurosurgery.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Clinical Dementia Rating (CDR) | pre treatment / ten days later (post treatment)
  The Clinical Dementia Rating is an assessment tool that primarily focuses on six domains: memory, orientation, judgment and problem-solving ability, community affairs, home and hobbies, and personal care. The questionnaire consists of two parts: the first part is answered by a caregiver and provides basic information about the individual (standard answers), while the second part is answered by the individual to compare against the answers from the first part. Each domain is scored from 0 to 3, with higher scores indicating more severe symptoms.
Mini-Mental State Examination (MMSE) | pre treatment / ten days later (post treatment)
  The MMSE consists of seven major domains: orientation, attention, memory, language, verbal comprehension, ability to perform tasks, and constructional ability. The total score is 30 points, with a cutoff typically set at 24 points; a score of 23 or lower indicates cognitive impairment.
Montreal Cognitive Assessment (MoCA): | pre treatment / ten days later (post treatment)
  The test consists of 30 points and takes 10 minutes for the individual to complete. The basics of this test include short-term memory, executive function, attention, focus, and more.
N-Back Test | pre treatment / ten days later (post treatment)
  The N-Back task is a series of stimuli that requires participants to respond when the current stimulus matches one presented n times before. In this study, a 2-Back test is used, meaning participants are asked to respond when they detect a stimulus that matches the one presented 2 stimuli ago.
Stroop Color Word Test (SWCT) | pre treatment / ten days later (post treatment)
  Also known as the Color-Word Conflict Test, it requires the individual to quickly read the color of the text (e.g., red, blue, green) rather than its meaning.
Wisconsin Card Sorting Test (WCST) | pre treatment / ten days later (post treatment)
  The WCST involves using four stimulus cards and a reference card. Participants are not informed of the pairing rules (color, shape, number form) and must choose a stimulus card to match with a response card. The tester provides feedback as "correct" or "incorrect." When the participant correctly pairs 10 cards in a row using the same rule, the tester changes the pairing rule. This test assesses the individual's executive function.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, New Taipei City, ROC, Taiwan

IPD SHARING:
Plan to Share IPD: No